CLINICAL TRIAL: NCT05135078
Title: Monitoring Risks for Hematological Changes in Gas Station Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Talaat Taha, Principal investigator ., Sohag University
Other Study IDs: Soh-Med-21-10-08
Record Dates: First submitted 2021-10-14; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gas station workers are exposed to carcinogenic substances.This increases risk of their exposure to hematological diseases such as lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL), myelodysplastic syndromes (MDS), and myelogenous leukemia (AML), as well as different forms of non-Hodgkin's lymphoma (NHL) and multiple myeloma. Thus, the early identification of this condition between the gas station workers may prevent the hematological disease progression.

DETAILED DESCRIPTION:
Gas station workers are exposed to carcinogenic substances.This increases risk of their exposure to hematological diseases such as lymphoblastic leukemia (ALL), chronic lymphocytic leukemia (CLL), myelodysplastic syndromes (MDS), and myelogenous leukemia (AML), as well as different forms of non-Hodgkin's lymphoma (NHL) and multiple myeloma.

It is known that severe bone marrow dysplasia is frequently accompanied by early alterations in the immune system and in peripheral cell subsets.

The bone marrow injury by benzene metabolites is a strong predisposing factor in the pathogenesis of Benzene-induced hematopoietic disease .Thus, the early identification of this condition between the gas station workers may prevent the hematological disease progression.

The reactive metabolite of benzene, 1,4-benzoquinone (BQ) is suggested to be a key molecule of benzene-induced hematotoxicity and carcinogenicity as it cause abnormal accumulation of myeloid cells and precursors, which cause benzene induced cytopenia and myeloid dysplasia in humans.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted on a group of gas station workers exposed to benzene for more than 3 years .

Exclusion Criteria:

* diagnosed gas station workers with blood malignancies .
* gas station workers exposed to benzene for less than 3 years .

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: gas station workers exposed to benzene more than 3 years
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The aim of study is to evaluate and monitor risks for hematological changes in gas station workers | within 6 months .
  The study will be conducted to a group of gas station workers exposed to benzene for more than 3 years, All workers will be subjected to complete blood count .
The aim of study is to evaluate and monitor risks for hematological changes in gas station workers | within 6 months .
  The study will be conducted to a group of gas station workers exposed to benzene for more than 3 years, All workers will be subjected to liver function tests as alanine transaminase (ALT) measured by IU/L, aspartate transaminase (AST) measured by IU/L, total protein measured by gm/dl, albumin measured by g/dl and bilirubin measured by mg/dl.
The aim of study is to evaluate and monitor risks for hematological changes in gas station workers | within 6 months .
  The study will be conducted to a group of gas station workers exposed to benzene for more than 3 years, All workers will be subjected to renal function tests as serum creatinine measured by mg/dl, serum urea measured by mg/dl and uric acid measured by mg/dl .
The aim of study is to evaluate and monitor risks for hematological changes in gas station workers | within 6 months .
  The study will be conducted to a group of gas station workers exposed to benzene for more than 3 years, All workers will be subjected to CD45, CD34, HLA-DR, CD33, CD13, CD19, CD22, CD2, CD3, CD5, CD7, CD4, CD8, CD10, CD16 and CD65 measured by flowcytometry
The aim of study is to evaluate and monitor risks for hematological changes in gas station workers | within 6 months ,
  The study will be conducted to a group of gas station workers exposed to benzene for more than 3 years, All workers will be subjected to ESR (Erythrocyte sedimentation rate) measured by mm .